CLINICAL TRIAL: NCT01193400
Title: Multicentric Phase II Trial, Prospective, Open, Single Group, to Discuss Induction Therapy With a Combination of Clofarabine and Low-dose Cytarabine Followed by Consolidation Therapy With Clofarabine and Low-dose Cytarabine for the Treatment of AML Patients Age Greater Than or Equal to 60 Years
Brief Title: Clofarabine and Low-dose Cytarabine Followed by Consolidation Therapy in AML Patients Age Greater Than or Equal to 60 Years
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Dr Miguel Angel Sanz, PETHEMA Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-CLOFARA-CA09; 2010-019718-25 (EudraCT Number)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute myelogenous leukemia; Clofarabine; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine-Cytarabine (Experimental): Induction therapy with a combination of clofarabine and low-dose cytarabine followed by consolidation therapy with clofarabine and low-dose cytarabine
  Interventions: Drug: Clofarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Clofarabine
Drug: Cytarabine

SUMMARY:
Primary outcome measure:

Evaluate the efficacy in terms of complete responses of induction therapy and first-line consolidation of Clofarabine and low-dose Cytarabine with AML patients aged 60 years or more. The first efficacy objective is evaluate the overall remission rate (TRG), where general reference (RG) is defined as a patient who achieved complete remission (CR) or complete remission with inadequate platelet recovery (CPR).

Secondary outcome measures:

* To evaluate disease-free survival (DFS)
* Evaluate the overall survival (OS)
* To evaluate the safety and tolerability of clofarabine and duration, severity and relationship of adverse events (AEs) occurring during treatment
* To assess the rate of mortality at 30 days (ie, the incidence of deaths occurring between Day 1 and Day 30 of induction cycle)
* The incidence, intensity (according to the latest version of the CTCAE classification), duration, causality, severity and type of AA

DETAILED DESCRIPTION:
This protocol corresponds to a multicenter, phase II, open, non randomized, designed to determine the efficacy of clofarabine and low-dose cytarabine combination in AML patients older than or equal to 60 years.

The trial is divided into pre-treatment and treatment (cycle / s of induction and consolidation) periods.The induction cycle consist of clofarabine at 20 mg/m2/day intravenously for 5 consecutive days plus cytarabine subcutaneously at 20 mg/m2/day for 14 consecutive days. If patients do not achieve CR they will receive a second course of induction with the same pattern. Consolidation cycles consist of clofarabine intravenously at 15 mg/m2/day for 5 consecutive days plus cytarabine at 20 mg/m2/day subcutaneously for 7 consecutive days. Patients will receive a maximum of 12 cycles of clofarabine and LDAC. The monitoring phase of survival is made by clinical practice and will continue until all patients have either died or survived two years after the end of treatment visit.

There will be 75 patients older than or equal to 60 years. Patients will be evaluated over the following periods: Pre-treatment and treatment (induction and consolidation).

Pre-treatment phase: includes enrolment visit in which the patient completes the written informed consent to participate in the study.

There will be a selection of patients who have given their written informed consent to join the clinical trial. They must meet all the inclusion criteria and no exclusion.

Treatment phase: Patients should begin treatment within 14 days after signing the informed consent form (ICF). Selection period begins when the ICF is signed and the inclusion period begins when the patient first receives the study drug (ie Day 1 of the induction cycle).

Safety will be evaluated by monitoring all adverse events haematological and not haematological related with the drug's study.

The final visit of treatment will take place at least 45 days after the last dose of study drug administration.

Patients who leave the study prematurely, should have the end of treatment visit within 2 weeks after the decision not to continue to administer the study drug. The final visit should take place within 2 weeks after the visit of the last cycle of treatment.

Off protocol, after making the final visit of, all patients receiving at least one dose of study drug will be subject to monitoring by normal clinical practice, for a minimum of two years from the final visit or until his death

Follow up phase:

The maximum follow-up for all patients is 2 years from the final visit of the last patient included and be conducted on a monthly basis during the first year and quarterly during the second at least, notwithstanding that there may be more visits at discretion of each centre or depending on the clinical features.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML (de novo, secondary, or hematological disorder), according to WHO criteria.
2. Older than or equal to 60 years
3. ECOG performance status 0-2
4. At least one of the following factors:

   * Older than or equal to 70 years
   * Prior hematological disorder (AHD)
   * ECOG performance status 2
   * Unfavorable karyotype (ie, adverse) defined as any cytogenetic profile except the presence of any of the following:

     t(8;21)(q22;q22) inv(16)(p13q22) or t(16;16)(p13;q22) t(15;17)(q22;q12) and variants
5. Provide written informed consent form.
6. Being able to comply with study procedures and follow-up evaluations.
7. Not to be fertile or willing to use a method of birth control during the study until the end of the last visit of the treatment.
8. Adequate renal and hepatic function as follows:

   * Total bilirubin <= 1,5 x upper of institutional normal limit (ULN) and
   * AST y ALT <=2,5 x ULN and
   * Serum creatinine <=1,0 mg/dL of serum creatinine <01,0 mg/dL, then, glomerular filtration rate (GFR) estimated must be >60 mL/min/1,73 m2 calculated from the equation of the Modification of Diet in Renal Disease (MDRD).
9. Adequate cardiac function determined by at least one of the following:

   * Left ventricular ejection fraction (LVEF) >=40% measured by echocardiography in Multiple Gated Acquisition (MUGA) scan or isotope angiography or
   * Left ventricular fractional shortening >=22% measured by echocardiography.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukaemia (APL) in French-American-British classification M3º or attending to the WHO classification t(15;17)(q22;q12), (PML/RAR and variants).
2. Pre-treatment with clofarabine.
3. Previous treatment for AML or a hematological disorder AHD (excluding palliative care, hydroxyurea, hematopoietic cytokines or lenalidomide [the latter only for a specific AHD]). Hematopoietic cytokines and lenalidomide should not have been administered within the 14 days preceding the first dose of study drug. If it is received any previous treatment for AML or AHD within the time limits allowed, drug-related toxicity, must have recovered to Grade 1 or less before the first dose of study drug.
4. Previous hematopoietic stem cell transplantation (HSCT).
5. External beam pelvic radiotherapy.
6. Have received an investigational product within 30 days before the first dose of study drug. If the patient has received any investigational product before this time, the drug-related toxicity, must have recovered to Grade 1 or less before the first dose of study drug.
7. Inadequate renal and hepatic function as follows:

   * Total bilirubin >1,5 x institutional upper limit normal (ULN) provided it is not attributable to the very LMA or
   * AST y ALT >2,5 x ULN provided it is not attributable to the very LMA or
   * Serum creatinine >1,0 mg/dL provided that the glomerular filtration rate (GFR) estimated to be ≤60 mL/min/1,73 m2 calculated by the equation of the Modification of Diet in Renal Disease (MDRD).
8. Inadequate cardiac function determined by at least one of the following:

   * Left ventricular ejection fraction <40% measured by echocardiography in Multiple Gated Acquisition (MUGA) or isotope angiography; or
   * Left ventricular fractional shortening <22% measured by echocardiography.
9. Poor general condition ECOG 3-4.
10. Refusal to sign informed consent form.
11. Inability to comply with study visits and inspections.
12. Psychiatric disorders that could interfere with the consent, participation or monitoring of the study.
13. Fungal Systemic disease, bacterial, viral or other uncontrolled infection (defined as manifestation of signs / symptoms related to ongoing infection and without improvement, although receiving adequate antibiotic therapy or other treatment).
14. Any other concomitant serious disease or a history of severe organ dysfunction or heart, kidney, liver or other organ system which may involve the patient in excessive risk when exposed to clofarabine.
15. Diagnosis of another malignancy neoplasia, unless the patient has been disease-free for at least five years after completing an attempt curative therapy with the following exceptions:

    * Patients with non-melanoma skin cancer, carcinoma in situ or cervical intraepithelial neoplasia, irrespective of the duration of disease-free period, are eligible for the study if it has finalized a definitive treatment for the disease.
    * Patients with prostate cancer confined to the organ without evidence of recurrent or progressive disease based on figures for the prostate specific antigen (PSA) are also candidates for the study if hormonal therapy has been initiated or has made a radical prostatectomy.
16. Clinical evidence which may indicate central nervous system (CNS) leukemia unless lumbar puncture to confirm the absence of leukemic blasts in the cerebrospinal fluid (CSF).
17. Previous positive test for human immunodeficiency virus (HIV).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 year
  Evaluate the efficacy in terms of complete responses of induction therapy and first-line consolidation of Clofarabine and low-dose Cytarabine with AML patients aged 60 years or more. The first efficacy objective is evaluate the overall remission rate (TRG), where general reference (RG) is defined as a patient who achieved complete remission (CR) or complete remission with inadequate platelet recovery (CPR).

SECONDARY OUTCOMES:
To evaluate disease-free survival (DFS)
Evaluate the overall survival (OS)
To evaluate the safety
To assess the rate of mortality at 30 days
• The incidence, intensity (according to the latest version of the CTCAE classification), duration, causality, severity and type of AE

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital Juan Canalejo., A Coruña
  - Hospital General de Alicante., Alicante
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital Durán i Reynals (Bellvitge)., Barcelona
  - Hospital Vall d' Hebron, Barcelona
  - ICO Hospital Germans Trias I Pujol., Barcelona
  - Hospital Reina Sofía., Córdoba
  - Hospital 12 de Octubre., Madrid
  - Hospital Ramón y Cajal., Madrid
  - Hospital San Pedro de Alcántara., Málaga
  - Hospital Central de Asturias., Oviedo
  - Hospital Clínico Universitario de Salamanca., Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valencia., Valencia
  - Hospital Universitario La Fe., Valencia

REFERENCES:
- [Derived] Martinez-Cuadron D, Montesinos P, Oriol A, Salamero O, Vidriales B, Bergua J, Herrera P, Vives S, Sanz J, Carpio C, Rodriguez-Veiga R, Moscardo F, Sanz MA. Phase II trial to assess the safety and efficacy of clofarabine in combination with low-dose cytarabine in elderly patients with acute myeloid leukemia. Ann Hematol. 2014 Jan;93(1):43-6. doi: 10.1007/s00277-013-1914-y. Epub 2013 Oct 1. PMID 24081577
- See also: Related Info — http://www.seif88.com